CLINICAL TRIAL: NCT02261441
Title: Identificación de la poBlación Española de RIesgo CArdiovascular y reNal
Brief Title: Cardiovascular and Renal Risk in Spain
Acronym: IBERICAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: La Sociedad Española de Médicos de Atención Primaria (Other)
Responsible Party: Principal Investigator, Carlos Escobar, MD, PhD, La Sociedad Española de Médicos de Atención Primaria
Other Study IDs: IBERICAN
Record Dates: First submitted 2014-09-27; First posted 2014-10-10 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Hypertension; Diabetes; Smoking; Hypercholesterolemia; Cardiovascular risk factor
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Smoking; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Subjects irrespective of the presence of risk factors or cardiovascular disease throughout Spain will be included. This is an observational and non-interventional study
  Interventions: Other: Observational and noninterventional study

INTERVENTIONS:
Other: Observational and noninterventional study — No specific recommendations will be provide to physicians about treatments. As a result, treatments of patients will be prescribed, modified or withdrawn according only to physicians´ judgment.

SUMMARY:
IBERICAN is a multicenter, longitudinal and observational population-based study of patients daily attended in Primary Care setting in Spain.

This study is aimed to determine the prevalence and incidence of cardiovascular risk factors in adult population in Spain.

Patients will be followed-up for a minimum period of 5 years, every 6 months or a lesser period when clinically required.

It has been estimated that a total of 15,000 individuals will be included.

DETAILED DESCRIPTION:
IBERICAN (Identificación de la poBlación Española de RIesgo CArdio Vascular y reNal) is a multicenter, longitudinal and observational population-based study of patients daily attended in Primary Care setting in Spain.

The aims of IBERICAN are to determine the prevalence and incidence of cardiovascular risk factors in adult population in Spain. Moreover, the development of cardiovascular outcomes, and risk factors control rates will be also analyzed.

In IBERICAN, subjects irrespective of the presence of risk factors or cardiovascular disease throughout Spain will be included.

No specific recommendations will be provide to physicians about treatments. As a result, treatments of patients will be prescribed, modified or withdrawn according only to physicians´ judgment. The study has been approved by the ethic committee of Hospital Carlos III, Madrid on February 2013. Before inclusion, every patient will provide a written informed consent.

Patients will be followed-up for a minimum period of 5 years, every 6 months or a lesser period when clinically required. Excepting a blood analysis in the previous 6 months before the inclusion, no other specific diagnostic tool or technique will be required for being included in the study. All blood and urine analysis or other techniques will be performed according to clinical practice during the follow-up.

It has been estimated that a total of 15,000 individuals will be included.

ELIGIBILITY:
Inclusion Criteria:

* National Health Care System user.
* Resident at Spain in the last 5 years.
* Attended by investigator in Primary Care setting.

Exclusion Criteria:

* Change of regular residence to other city or country in the following 6 months.
* Life expectancy less than 5 years.
* Difficult to follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects irrespective of the presence of risk factors or cardiovascular disease throughout Spain
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular event | 5 years
  Development of cardiovascular events.
Cardiovascular risk factors | 5 years
  Development of cardiovascular risk factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Goya, 25, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cavelaars AE, Kunst AE, Geurts JJ, Crialesi R, Grotvedt L, Helmert U, Lahelma E, Lundberg O, Matheson J, Mielck A, Mizrahi A, Mizrahi A, Rasmussen NK, Regidor E, Spuhler T, Mackenbach JP. Differences in self reported morbidity by educational level: a comparison of 11 western European countries. J Epidemiol Community Health. 1998 Apr;52(4):219-27. doi: 10.1136/jech.52.4.219. PMID 9616407
- [Result] Marrugat J, Elosua R, Marti H. [Epidemiology of ischaemic heart disease in Spain: estimation of the number of cases and trends from 1997 to 2005]. Rev Esp Cardiol. 2002 Apr;55(4):337-46. doi: 10.1016/s0300-8932(02)76611-6. Spanish. PMID 11975899
- [Result] Fiol M, Cabades A, Sala J, Marrugat J, Elosua R, Vega G, Jose Tormo Diaz M, Segura A, Aldasoro E, Moreno-Iribas C, Muniz J, Hurtado de Saracho I, Garcia J. [Variability in the in-hospital management of acute myocardial infarction in Spain. IBERICA Study (Investigacion, Busqueda Especifica y Registro de Isquemia Coronaria Aguda)]. Rev Esp Cardiol. 2001 Apr;54(4):443-52. doi: 10.1016/s0300-8932(01)76332-4. Spanish. PMID 11282049
- [Result] Marrugat J, Sanz G, Masia R, Valle V, Molina L, Cardona M, Sala J, Seres L, Szescielinski L, Albert X, Lupon J, Alonso J. Six-month outcome in patients with myocardial infarction initially admitted to tertiary and nontertiary hospitals. RESCATE Investigators. Recursos Empleados en el Sindrome Coronario Agudo y Tiempos de Espera. J Am Coll Cardiol. 1997 Nov 1;30(5):1187-92. doi: 10.1016/s0735-1097(97)00312-4. PMID 9350913
- [Result] Gispert Magarolas R, Bares Marcano MA, Freitas Ramirez A, Torne Farre M, Puigdefabregas Serra A, Alberquilla A, Albert X, Luis Alfonso J, Caminal J, Fernandez-Cuenca R, Garcia F, Gervas J, Librero J, Martos C, Medrano MJ, Ruiz M. [Health system interventions assessment in Spain: an approach through the analysis of the time trends and the geographical variability of avoidable mortality between 1986 -2001]. Rev Esp Salud Publica. 2006 Mar-Apr;80(2):139-55. doi: 10.1590/s1135-57272006000200004. Spanish. PMID 16719023
- [Result] Felix-Redondo FJ, Fernandez-Berges D, Grau M, Baena-Diez JM, Mostaza JM, Vila J. Prevalence and clinical characteristics of peripheral arterial disease in the study population Hermex. Rev Esp Cardiol (Engl Ed). 2012 Aug;65(8):726-33. doi: 10.1016/j.recesp.2012.03.008. Epub 2012 Jun 22. English, Spanish. PMID 22727799
- [Result] Daniels SR. Prevention of atherosclerotic cardiovascular disease: what is the best approach and how early should we start? J Am Coll Cardiol. 2014 Jul 1;63(25 Pt A):2786-8. doi: 10.1016/j.jacc.2014.01.082. Epub 2014 May 7. No abstract available. PMID 24814499
- [Result] Persic V. Obesity in the cardiovascular continuum. Curr Clin Pharmacol. 2013 May;8(2):159-63. doi: 10.2174/1574884711308020008. PMID 22950957
- [Result] Burgmaier M, Heinrich C, Marx N. Cardiovascular effects of GLP-1 and GLP-1-based therapies: implications for the cardiovascular continuum in diabetes? Diabet Med. 2013 Mar;30(3):289-99. doi: 10.1111/j.1464-5491.2012.03746.x. PMID 22804451
- [Result] Gonzalez-Juanatey JR, Cordero A. Benefits of delapril in hypertensive patients along the cardiovascular continuum. Expert Rev Cardiovasc Ther. 2013 Mar;11(3):271-81. doi: 10.1586/erc.12.188. PMID 23469905
- [Result] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213
- [Result] Bastuji-Garin S, Deverly A, Moyse D, Castaigne A, Mancia G, de Leeuw PW, Ruilope LM, Rosenthal T, Chatellier G; Intervention as a Goal in Hypertension Treatment Study Group. The Framingham prediction rule is not valid in a European population of treated hypertensive patients. J Hypertens. 2002 Oct;20(10):1973-80. doi: 10.1097/00004872-200210000-00016. PMID 12359975
- [Result] Marrugat J, Subirana I, Comin E, Cabezas C, Vila J, Elosua R, Nam BH, Ramos R, Sala J, Solanas P, Cordon F, Gene-Badia J, D'Agostino RB; VERIFICA Investigators. Validity of an adaptation of the Framingham cardiovascular risk function: the VERIFICA Study. J Epidemiol Community Health. 2007 Jan;61(1):40-7. doi: 10.1136/jech.2005.038505. PMID 17183014
- [Result] Mazon-Ramos P. [Cardiovascular risk in the 21st century: identifying risk in primary prevention. Controlling risk in secondary prevention]. Rev Esp Cardiol (Engl Ed). 2012 Jul;65 Suppl 2:3-9. doi: 10.1016/j.recesp.2012.07.004. Spanish. PMID 22921168
- [Result] Kavouras SA, Panagiotakos DB, Pitsavos C, Chrysohoou C, Arnaoutis G, Skoumas Y, Stefanadis C. Physical Activity and Adherence to Mediterranean Diet Increase Total Antioxidant Capacity: The ATTICA Study. Cardiol Res Pract. 2010 Oct 20;2011:248626. doi: 10.4061/2011/248626. PMID 20981278
- [Result] Panagiotakos DB, Pitsavos C, Stefanadis C. Dietary patterns: a Mediterranean diet score and its relation to clinical and biological markers of cardiovascular disease risk. Nutr Metab Cardiovasc Dis. 2006 Dec;16(8):559-68. doi: 10.1016/j.numecd.2005.08.006. Epub 2006 Feb 9. PMID 17126772
- [Derived] Cinza-Sanjurjo S, Prieto-Diaz MA, Pallares-Carratala V, Mico-Perez RM, Velilla-Zancada S, Barquilla-Garcia A, Ginel-Mendoza L, Segura-Fragoso A, Martin-Sanchez V, Polo-Garcia J. Characteristics of the phenotypes in prevalent and incident cases of heart failure in primary care: IBERICAN study. BMC Prim Care. 2024 Jul 25;25(1):271. doi: 10.1186/s12875-024-02506-1. PMID 39054420